CLINICAL TRIAL: NCT04587921
Title: Feasibility and Impact of Remote Oximetry and Cardiac Frequency Monitoring in Patients Hospitalized and Isolated With Covid-19
Brief Title: Feasibility and Impact of Remote Oximetry in Patients Hospitalized With Covid-19
Acronym: MoxiCov
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Associate Professor/PI, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5058/20/087
Record Dates: First submitted 2020-08-18; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Oximetry; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients monitored with oximeter (Experimental): The first 45 patients will be monitored but the results will not be displayed. The second half of the patients the oximeter will have their monitoring data available online in the ward.
  Interventions: Device: Digital oximeter monitoring

INTERVENTIONS:
Device: Digital oximeter monitoring — Digital oximeter and cardiac frequency monitoring.

SUMMARY:
The objective of MoxiCov is to monitor the oximetry of patients admitted to the Covid nursery to provide a more detailed assistance expecting to reduce the amount of hypoxia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* COVID 19 positive or suspected COVID19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-06-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the system: Determination of the number of valid versus not valid or missed measurements | 6 months
  Determination of the number of valid versus not valid or missed measurements of each participant.
Hypoxic burden | 6 months
  Time spent with SpO2< 93%, 90% and 85%
Hypoxic alarm | 6 months
  Number of times the oximeter record 3 consecutive measurements of SpO2<90%
Satisfaction of the nursing, medical team and patients with the implemented system | 6 months
  Measurement of NET PROMOTING SCORE (NPS). This score will show the satisfaction of the healthcare team with the device. This score have a minimum of 0 points and maximum of 32 points.

SECONDARY OUTCOMES:
Time of SpO2<90%, SpO2<85% and SpO2<80% | 6 months
Number of false alarms caused by malfunctions or bad oximeter positioning | 6 months
Total hospital stay | 6 months
Time of supplementary oxygen use | 6 months
Mortality of participants | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fundação Zerbini - Instituto do Coração (InCor), São Paulo, São Paulo, Brazil